CLINICAL TRIAL: NCT03581812
Title: Snack Foods and Their Impact on Gastrointestinal Physiology, Luminal Microbiology and Gastrointestinal Symptoms
Brief Title: Snack Foods and Their Impact on Gastrointestinal Microbiology, Function and Symptoms
Acronym: OptiGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Queen Mary University of London (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Professor Kevin Whelan, Professor of Dietetics, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HR-17/18-5341
Record Dates: First submitted 2018-06-23; First posted 2018-07-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Human Microbiome; Eating Behavior
Keywords: Gut Microbiota; Microbiome; Gut Health; Snack
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention snack 1 (Active Comparator): Snack food believed to selectively promote the growth of beneficial bacterial strains in the human colon.
  Interventions: Dietary Supplement: Intervention snack 1
- Intervention snack 2 (Active Comparator): Snack food believed to selectively promote the growth of beneficial bacterial strains in the human colon.
  Interventions: Dietary Supplement: Intervention snack 2
- Control snack (Placebo Comparator): Control snack food reflecting the macro-nutrient profile of a typical UK snack.
  Interventions: Dietary Supplement: Control snack

INTERVENTIONS:
Dietary Supplement: Intervention snack 1 — To be eaten instead of regular snacks twice a day for 4 weeks.
  Arms: Intervention snack 1
Dietary Supplement: Intervention snack 2 — To be eaten instead of regular snacks twice a day for 4 weeks.
  Arms: Intervention snack 2
Dietary Supplement: Control snack — To be eaten instead of regular snacks twice a day for 4 weeks.
  Arms: Control snack

SUMMARY:
The purpose of this study is to evaluate the impact of replacing usual snacks with alternative snack foods on gut health in a population of habitual snackers with low fibre intake.

DETAILED DESCRIPTION:
Diet is a crucial target for the improvement of human health. In the modern world, diets are diverse and diet related diseases are becoming more and more common. In particular, it is becoming increasingly apparent that the bacteria that live in the gut are strongly linked to both diet and health. Bacteria in the gut can be beneficial or harmful, and the health of the gut relies on the beneficial bacteria outnumbering the harmful ones. Diet has a great impact on the bacterial composition of the gut. In turn, the gut bacteria play diverse roles in human health, influencing not only the gut but also the health of the immune system, heart and brain. Therefore, optimising the composition of the gut bacterial is vital to human health and wellbeing.

It has been shown that snacks between meals contributes 420 - 480 calories per day, almost a quarter of the recommended intake. Therefore, snack choices are an area of diet and lifestyle that have the potential to influence diet and in turn the health of our gut and gut bacteria. We would like to assess the effect of replacing usual snacks with alternative snack foods that we believe have benefits for gut health.

The primary aim of the study is to investigate whether the replacement of usual snacks has an effect on gut bacterial composition, specifically the abundance of Bifidobacteria. Secondary aims include the effect of the intervention snacks on additional measures of gut health such as gut transit time, the frequency and consistency of bowel movements and gut symptoms e.g. heartburn, nausea, belching etc. The effect of snack foods on metabolites in the blood (e.g. glucose, insulin, lipids) will also be determined. Finally the impact of snack replacement on mood and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 18-45 years
* Body mass index (BMI) of 18.5 - 29.9 kg/m2
* Regular consumption of snacks (≥2 per day, excluding fruit and nut snacks)
* Low fibre intake (<22 g/d)
* Willing to follow the protocol and provide consent

Exclusion Criteria:

* Allergy or intolerance to snack ingredients (assessed at screening)
* Dislike of study snacks
* Regular consumption of intervention foods as snacks (twice a day in last month)
* Diabetes
* Major active psychiatric conditions (e.g. schizophrenia) or current eating disorder
* Active treatment for cancer in the last year
* Severe renal, cardiac or pulmonary disease or any other chronic medical condition
* Severe oesophagitis, gastritis or duodenitis
* Active diverticulitis or intestinal/colonic strictures
* Crohns disease or Ulcerative colitis
* Abdominal surgery (except appendicectomy or cholecystectomy)
* Irritable bowel syndrome
* Functional constipation
* Functional diarrhoea
* Antibiotics (past 4 weeks)
* Ongoing therapy with drugs affecting gastrointestinal motility
* Use of medical devices (Pacemakers, infusion pumps, insulin pumps)
* Women who are pregnant/lactating/planning pregnancy
* Recent/ongoing consumption of probiotics/prebiotics (past 4 weeks)
* Ongoing abuse of alcohol/drugs/other medication
* Very high physical activity levels
* Unexplained/unintentional weight loss in the past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Faecal bifidobacteria | Baseline
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from participant stool samples
Faecal bifidobacteria | Day 28
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from participant stool samples

SECONDARY OUTCOMES:
Whole gut transit time | Baseline
  Measured using the SmartPill wireless motility capsule
Whole gut transit time | Day 28
  Measured using the SmartPill wireless motility capsule
Regional gut transit time | Baseline
  Measured using the SmartPill wireless motility capsule
Regional gut transit time | Day 28
  Measured using the SmartPill wireless motility capsule
Regional gut pH | Baseline
  Measured using the SmartPill wireless motility capsule
Regional gut pH | Day 28
  Measured using the SmartPill wireless motility capsule
Faecal gut microbiota (alpha- and beta-diversity) | Baseline
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from participant stool samples
Faecal gut microbiota (alpha- and beta-diversity) | Day 28
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from participant stool samples
Faecal short-chain fatty acids (SCFA) | Baseline
  Measured by gas liquid chromatography of stool sample
Faecal short-chain fatty acids (SCFA) | Day 28
  Measured by gas liquid chromatography of stool sample
Faecal water | Baseline
  Measured by lyophilization of stool sample
Faecal water | Day 28
  Measured by lyophilization of stool sample
Faecal volatile organic compounds | Baseline
  Measured by gas-chromatography mass-spectrometry of stool samples
Faecal volatile organic compounds | Day 28
  Measured by gas-chromatography mass-spectrometry of stool samples
Gut symptoms | Week 0
  Gastrointestinal symptoms rating scale (7-day; questionnaire)
Gut symptoms | week 4
  Gastrointestinal symptoms rating scale (7-day; questionnaire)
Stool frequency | Week 0
  Bristol stool form scale (7-day; questionnaire)
Stool frequency | Week 4
  Bristol stool form scale(7-day; questionnaire)
Dietary intake | Week 0
  7-day food diary
Dietary intake | Week 4
  7-day food diary
Quality of life | Baseline
  SF-36 questionnaire
Quality of life | Day 28
  SF-36 questionnaire
Mood | Baseline
  Hospital anxiety and depression scale
Mood | Day 28
  Hospital anxiety and depression scale
Physical activity | Baseline
  Recent physical activity questionnaire
Physical activity | Day 28
  Recent physical activity questionnaire
Dietary metabolites (various) | Baseline
  Measured in blood sample
Dietary metabolites (various) | Day 28
  Measured in blood sample
Particle size of masticated snack foods | Day 28
  Mechanical sieving and laser diffraction of masticated snack foods

OTHER OUTCOMES:
Adverse events | From baseline - day 28
  Interview-administered questionnaire
Acceptability of snack products | Day 28
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Whelan, Prof., Principal Investigator — King's College London
Locations (1):
- King's College London Waterloo Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creedon AC, Dimidi E, Hung ES, Rossi M, Probert C, Grassby T, Miguens-Blanco J, Marchesi JR, Scott SM, Berry SE, Whelan K. The impact of almonds and almond processing on gastrointestinal physiology, luminal microbiology, and gastrointestinal symptoms: a randomized controlled trial and mastication study. Am J Clin Nutr. 2022 Dec 19;116(6):1790-1804. doi: 10.1093/ajcn/nqac265. PMID 36130222